CLINICAL TRIAL: NCT07354373
Title: The Efficacy of Single-Visit and Two-Visit Endodontic Treatments for Necrotic Teeth With Apical Periodontitis
Brief Title: Single-Visit and Two-Visit Endodontic Treatments
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ucsfendo
Record Dates: First submitted 2025-12-05; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Endodontic Infection; Periapical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis | interventions — Calcium Hydroxide; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-visit endodontic treatment (Experimental): In this arm, obturation will be completed using a single-cone technique after cleaning and shaping.
  Interventions: Other: control group
- multiple visits endodontic treatment (Experimental): in this arm the endodontic therapy will be completed in multiple visits.
  Interventions: Other: Calcium Hydroxide (CH)

INTERVENTIONS:
Other: Calcium Hydroxide (CH) — calcium hydroxide will be used as interim medication in the first visit and patients will return for the obturation in the second visit.
  Arms: multiple visits endodontic treatment
Other: control group — control group- no intervention
  Arms: One-visit endodontic treatment

SUMMARY:
You are being asked to participate in this research study because you are being treated at the UCSF Graduate Endodontics department for an endodontic procedure. We are trying to determine the treatment outcomes of one v. two-visit endodontic treatments. .If you decide to continue, we would like to request your consent for a follow up period of 1 year to observe the healing of the abscess. Observation periods occur at 6 months following the completion of the root canal and at 12 months and are a part of the standard of care. We will review findings in the Axium chart, which will be recorded by the treating doctor

DETAILED DESCRIPTION:
This research study includes patients who are receiving endodontic treatment within the UCSF Graduate Endodontics Department. The purpose of the study is to evaluate and compare treatment outcomes between one-visit and two-visit root canal procedures. Participants who choose to continue in the study will be followed for a period of one year so that healing of the periapical abscess can be monitored. Follow-up appointments are scheduled at six months and twelve months after treatment completion, both of which are part of routine standard care. Clinical and radiographic findings documented in the Axium chart by the treating provider will be reviewed as part of the study analysis.

ELIGIBILITY:
Inclusion Criteria:

* Classified as American Society of Anesthesiologists (ASA) Class I or II
* presenting with radiographic evidence of apical periodontitis-defined as a Cone-Beam Computed Tomography Periapical Index (CBCTPAI) score of 3 or greater according to the Estrela classification

Exclusion Criteria:

* Exclusion criteria included patients with uncontrolled chronic systemic conditions (e.g., diabetes, hypertension, chronic obstructive pulmonary disease), cardiovascular disease, renal or hepatic impairment, and autoimmune disorders
* History of smoking
* Periodontal disease with probing depths ≥ 3 mm.
* Root fractures
* Immature apices
* Resorption
* perforations
* Inability to achieve rubber dam isolation
* Lack of informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Clinical and Radiographic Healing | 12 months
  The primary outcome was defined using a combined clinical and radiographic healing based on the Cone-Beam Computed Tomography Periapical Index (CBCT-PAI)

SECONDARY OUTCOMES:
Volumetric Change in Periapical Lesion Size | 12 months
  The secondary outcome was defined as the change in lesion volume (mm³) between baseline and follow-up CBCT scans, serving as a quantitative metric of periapical healing

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Francisco School of dentistry, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Siqueira JF Jr, Rôças IN. Clinical implications and microbiology of bacterial persistence after treatment procedures. J Endod 2008;34:1291-1301. 2. Tait C, Camilleri J, Blundell K. Non-surgical endodontics: obturation. Br Dent J 2025;238:487-496. 3. Schwendicke F, Göstemeyer G. Cost-effectiveness of single- versus multistep root canal treatment. J Endod 2016;42:1446-1452. 4. Makanjuola JO, Umesi DC, Oderinu OH. Comparison of the incidence of flare-up and time efficiency in single-visit root canal treatment employing either rotary or manual step-back canal preparatory technique. Niger Postgrad Med J 2018;25:100-104. 5. Ricucci D, Siqueira JF Jr. Biofilms and apical periodontitis: prevalence and association with clinical and histopathologic findings. J Endod 2010;36:1277-1288. 6. Siqueira JF Jr. Reaction of periradicular tissues to root canal treatment: benefits and drawbacks. Endod Topics 2005;10:123-147. 7. Shuping GB, Ørstavik D, Sigurdsson A, Trope M. Reduction of intracanal bacteria using nickel-titanium rotary instrumentation and various medications. J Endod 2000;26:751-755. 8. Sjögren U, Figdor D, Spångberg L, Sundqvist G. The antimicrobial effect of calcium hydroxide as a short-term intracanal dressing. Int Endod J 1991;24:119-125. 9. Tronstad L, Andreasen JO, Hasselgren G, et al. pH changes in dental tissues after root canal filling with calcium hydroxide. J Endod 1981;7:17-21. 10. Ng YL, Mann V, Rahbaran S, et al. Outcome of primary root canal treatment: systematic review-Part 2. Influence of clinical factors. Int Endod J 2008;41:6-31. 11. Mergoni G, Ganim M, Lodi G, et al. Single versus multiple visits for endodontic treatment of permanent teeth. Cochrane Database Syst Rev 2022;12:CD004450. 12. Schulz KF, Altman DG, Moher D. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. J Pharmacol Pharmacother 2010;1:100-107. 13. Estrela C, Bueno MR, Azevedo BC, et al. A new periapical index based on cone-beam computed tomogr